# A Real-world Clinical Study on the Treatment of Menopausal Syndrome With Liuwei Dihuang Pills

**Informed Consent Form** 

2025.01.23

# Dear Mr. / Madam,

We would like to invite you to participate in a clinical study on "A Real-world Clinical Study on the Treatment of Menopausal Syndrome With Liuwei Dihuang Pills ."

Before you decide whether to participate in the study, read the following as carefully as possible. It will help you understand the study and why the study, the procedures and duration of the study, the benefits, risks and discomfort that may bring to you after participating in this study. If you wish, you can also discuss it with your relatives and friends, or ask your doctor to give an explanation to help you make a decision.

# Research introduction

#### —, Research background and study objectives

#### 1.research background

Menopause syndrome is a series of symptoms of autonomic dysfunction due to a decline in sex hormones before and after menopause. Often accompanied by menstrual cycle disorders, hot flushes, night sweats, sleep disorders, mood disorders and other neuropsychological symptoms. The core reason lies in the gradual decline of ovarian function, including natural menopause and artificial menopause. Due to the irreversible low-level estrogen status, postmenopausal aging lasts

for at least 30-40 years, which occupies ½ even longer, during which the incidence of complications also has increased significantly. About 25 million women worldwide enter menopause every year, and 10 million women in China enter menopause every year. The United Nations World Health Organization estimates that by 2030, the population of menopausal women worldwide will reach more than 1.2 billion, and the number of menopausal women in China will exceed 210 million, accounting for about 1 / 7 of the total population, which needs to be valued by public health.

The western medicine treatment of menopausal syndrome mainly focuses on psychological therapy and hormone therapy, but hormone supplementation often leads to diseases of other organs, such as breast cancer, cervical cancer, etc., which has certain limitations. Treatment of traditional Chinese medicine menopausal syndrome has thousands of years of history, menopausal syndrome in traditional Chinese medicine called "before and after the disease", belongs to the "lily disease", "dirty manic" category, the pathogenesis of the disease of the basic pathogenesis for menopause before and after the female kidney qi failure, decyl day, kidney imbalance of Yin and Yang, is the key to the syndrome before and after the menopause. The imbalance of Yin and Yang in the kidney often involves other viscera, mainly in the heart, liver and spleen. If the kidney Yin is insufficient and can not help the heart fire, the heart fire is high; the same, kidney Yin deficiency, kidney Yin deficiency, liver deficiency, liver flexibility, liver Yang hyperactivity; kidney and spleen days, kidney Yang warm, kidney deficiency Yang decay, the fire is not warm soil, and often cause spleen kidney Yang deficiency, water, the dampness, phlegm, blood stasis, depression, thus complex pathological mechanisms and various clinical symptoms.

Liuwei Dihuang Pills were first recorded in the "Direct Formula of Children", which is a

classic prescription for tonifying kidney, and was listed as the first batch of "Ancient Classic prescriptions" by the State Administration of Traditional Chinese Medicine. The prescription is composed of six traditional Chinese medicines, namely rehmannia, cornwood, peony skin, yam, poria cocos and Ze diarrhea. It has the effect of nourishing Yin and tonifying kidney. It is suitable for kidney Yin loss, dizziness and tinnitus, tenderness in waist and knee, bone steaming, night sweat and sperm and thirst elimination. Compound powder, nourishing Yin and tonifying kidney, tuckahoe removing dampness and invigorating the spleen, Chinese yam nourishing the spleen and kidney, nourishing the liver and kidney, and reducing the heat of the peony peel. It enhances immunity, reduces blood lipid, blood pressure, blood sugar, anti-fatigue, aging, low temperature, and resistance to hypoxia to improve kidney function, plant nervous system function, and has a promoting effect on metabolism. It can improve the estrogen level of menopausal women, promote the feedback control of the hypothalamic-pituitary-ovarian axis, improve the endocrine function and the internal environment of the body, and reduce the clinical symptoms. Traditional Chinese medicine treatment of menopausal syndrome from syndrome differentiation has distinct characteristics and advantages. Clinical observation and research have proved that TCM treatment of menopausal syndrome has definite effect and good safety.

Studies have shown that Liuwei Dihuang Pills combined with western medicine can treat hyperthyroidism and kidney Yin deficiency disease in children, and regulate the corresponding serum free triiodothyronine (FT3), free thyroxine (FT4) and thyroid stimulating hormone (TSH) levels. Sex hormone and thyroid hormone are governed by the thalamic-pituitary axis, and at the same time, thyroid hormone can improve the secretion of sex hormones, and sex hormones and thyroid hormones influence each other. Thyroid hormone plays an important auxiliary role in the regulation of sex hormones. Therefore, the abnormal secretion of thyroid gland aggravates the clinical symptoms of patients. In addition, there are few clinical studies on thyroid hormone and glucose and lipid metabolism in perimenopausal women, so further research is needed. The immune system is an indispensable defense system of the human body, and it plays a very important role in menopause. Studies have shown that the immune system of the human body is closely related to the neuroendocrine system. With the arrival of menopause, the neuroendocrine system of women is chaotic and its disease resistance gradually decreases. The ratio of CD4 / CD8 in T lymphocyte subsets reflects the human immune function. And the ratio of T cell subsets in the peripheral blood of healthy adults is between 1.5 and 2.0. With the decline of immune function of menopausal women, the composition, efficacy and transmission pathway of T cell subsets are change, mainly manifested as a drop of CD4 and CD8T cells. As a pleiotropic cytokine produced by a variety of cells, IL-6 mainly participates in the inflammatory response and immune response of the human body through humoral immunity. In the normal immune state, most of them are in the "dormant" state. With the decline of the body's immune function, the serum content of IL-6 increases significantly to enhance the ability to remove foreign foreign body antigen.

## 2 .Introduction to the study drug

Name: Liuwei Dihuang Pills.

Ingredients: cooked rehmannia, wine wood meat, peony skin, yam, poria cocos, diarrhea.

Character: this product is brown to black brown honey pill; sweet and sour taste.

Indications: nourishing the Yin and tonifying the kidney. For kidney Yin loss, dizziness and tinnitus, waist and knee sour and soft, bone steaming hot flashes, night sweat spermatorrhea.

Usage and dosage: Use drugs according to the instructions.

Specification: No limit.

Storage: seal.

This study belongs to the National Key Research and Development Program of Traditional Chinese Medicine modernization "Demonstration Study of clinical Efficacy and Safety Evaluation of proprietary Chinese Medicine based on Systems Biology"

(No.2022YFC3502004), funded by the project " Clinical Verification and Safety of Efficacy and Biomarker Discovery of proprietary Chinese patent Medicine". This research project was reviewed by the Ethics Committee of Beijing Longfu Hospital in accordance with the ethical principles of protecting the interests of relevant national regulations of China and the Declaration of Helsinki.

#### **\_\_\_\_\_**, Inclusion criteria, exclusion criteria, and discontinuation criteria

#### 1. Selection criteria:

- (1) Age: 45-55 years old (including both ends); Gender: female;
- (2) Meet the western medicine diagnostic criteria for menopausal syndrome;
- (3) Meet the TCM syndrome differentiation standard of kidney and Yin deficiency syndrome;
- (4) Informed consent, and the voluntary signing of the informed consent form.

#### 2. Exclusion criteria:

- (1) Those allergic to the ingredients and excipients;
- (2) Other endocrine diseases;
- (3)The presence of the reproductive system organic lesions;
- (4) Patients with bilateral oophorectomy, hysterectomy, and ovarian dysfunction;
- (5) Patients with endometrial hyperplasia, unexplained vaginal bleeding;
- (6) Patients with malignant tumors, hematopoietic system and immune system diseases;
- (7) Serious diseases of cardiovascular and cerebrovascular diseases, liver and kidney organs (serum transaminase level is more than 1.5 times higher than the upper limit of normal value, and serum creatinine is higher than the upper limit of normal value);
- (8) Psychiatric illness and alcohol or drug dependence;
- (9) With mental illness or communication disorder;
- (10) According to the judgment of the investigator, other lesions that reduce the possibility of enrollment or complicate the enrollment are not suitable to participate in this clinical study;

#### 3.Stop the standard

- (1) with serious adverse events or serious adverse reactions;
- (2) Request withdrawal from the investigator;
- (3) Patients with serious complications or other serious diseases who occurred during the study.

# **\equiv**, What will you need to do if you participate in the study?

1. If you meet the inclusion criteria and agree to participate, the study will follow the following steps:

Screening period (-14 to 0 days): as judged by the scale. Enrollment period (0 days): ①

Determine formal enrollment: subjects who meet the inclusion criteria, complete safety indicators and observation indicators are the qualified cases; ② Complete the CRF; ③ According to the doctor's prescription and the patient's own wishes (no drug is provided in this project); ④ pecify the date of next follow-up. One follow-up period (14±2 days): ① Adverse events and concomitant medication records; ② Determines the date of next follow-up; ③ To complete the CRF. The second follow-up period (28±2 days): ① Blood sampling test; ② To complete the CRF.

2. Other matters that require your cooperation: return a visit on time, report the improvement of symptoms and collect blood at the required time point.

## 四、Benefits from participating in the study

Participate in this clinical study, your condition may improve;

You can obtain the free examination, condition counseling service, and feedback group test results related to the study (see the protocol for details);

Your participation will also contribute to the real world clinical study of the treatment of menopausal syndrome, which is of social significance for the treatment of this disease and for other patients with such diseases.

# 五、Risk of participating in the study

In this study, about 6.5ml of blood will be collected before and after medication, and there may be some very small risks when the blood sampling, including temporary pain, local blue, and a few people will have mild dizziness. If you feel unwell during the study, tell your study physician immediately that he / she will judge and treat your discomfort.

#### 六、Expenses, compensation and compensation for participating in the study

Participating in this study will provide relevant laboratory tests, condition consultation services, and feedback of group test results free of charge.

If you do have any injury related to this study, the Sponsor / research group will be liable in accordance with national laws and regulations and provide corresponding compensation or compensation for the damage related to the trial.

If you combine the treatment and examination required for other diseases, it will not be free of charge.

#### 七、Is the personal information kept confidential?

Information about your participation in this study will be recorded in the study medical chart /case report form. All study findings (including personal data, laboratory documents, etc.) appearing in the original medical records will be kept completely confidential to the extent

permitted by law. Your name will not appear in the CRF table, only with your name pinyin abbreviation and the number assigned when you participate in the study. Related research summaries, articles, public publications, if necessary, will only appear your name pinyin abbreviation and number.

If necessary, the drug regulatory department, the ethics committee or the project funding department may consult the information of the subjects participating in the study. However, without permission, they will not use the subject data for other purposes or disclose it to other groups.

# 八、How do you get more information?

You can ask any questions about this study at any time.

Your doctor will leave you his / her phone number so you can answer your questions.

Your doctor will promptly notify you if there is any important new information during the study that may affect your willingness to continue participating in the study.

# 九、You can voluntarily choose to participate in the study and withdraw from the study midway

Participation in this study depends entirely on your willingness. You may refuse to participate in this study or withdraw from the study at any time during the study. If you opt out of this study, your benefits will not be affected and discriminated or retaliation.

Your doctor or investigator may suspend your participation in this study at any time for your best interest.

If you withdraw from the study for any reason, you may be consulted about your use of the study drug. You may also be required to have a laboratory and physical examination if your doctor considers it. You can also refuse without any discrimination or retaliation.

If you choose to participate in this study, we expect you to follow through the whole process.

#### +, What should I do now?

You will decide whether to participate in this study. You can discuss it with your family or friends before making a decision.

Before you make your decision to participate in the study, please ask your doctor any questions until you fully understand the study.

#### +-. The Ethics Committee

If you have any questions or need to ask anyone other than the investigator, please consult the Ethics Committee of Beijing Longfu Hospital.

The Office of the Ethics Committee:Science and Education Department of Beijing Longfu Hospital

Contact number:87947345

Thank you for reading the above materials. If you decide to participate in this study, please

tell your doctor that he  $\/$  she will arrange for the study.

Please keep this information.

# **Informed Consent consent signature page**

Project name: A Real-world Clinical Study on the Treatment of Menopausal Syndrome With Liuwei Dihuang Pills

Project source:"Research on Modernization of Traditional Chinese Medicine" of China (2022YFC3502004)

#### **Consent statement**

I have read the above introduction to this study and have the opportunity to discuss and ask questions about this study.

All the questions I have raised have been answered satisfactorily.

I am aware of the risks and benefits that may arise from participating in this study. I know that participation in the study is voluntary, and I confirm that I have enough time to consider it and understand that:

- ·I can consult my doctor for more information.
- ·I can withdraw from this study at any time without discrimination or retaliation, and my medical treatment and interests will not be affected.

I am also aware that if I withdraw from the study, especially due to drug reasons, if I tell the doctor about the changes in my condition and complete the corresponding physical examination and physical examination, it will be very beneficial to me and the whole study.

If any other medication is needed for the illness, I will ask the doctor for advice in advance or tell him the truth afterwards.

I agree with the representatives of the drug administration department, the ethics committee or the project funding department to access my research materials.

I will obtain a copy of the signed and dated informed consent form.

Finally, I decided to agree to participate in this study, and I promised to follow the doctor's advice as much as possible.

| | Subjects signed: | |
|---|---|---|
| | | Date: year, month, month and day |
| | Subject Contact Number: | |
| expl | I confirm that the details of the study including its rights and possible benefits and risks were explained to the subject and I give a copy of the signed informed consent form. | |

Investigator's signature:

Date: year, month, month and day

**Investigator Contact Number:**